CLINICAL TRIAL: NCT04014309
Title: Supportive and Survivorship Care Program for Cancer Patients: a Cluster Randomized Controlled Pilot Study Among Breast and Gynaecological Cancer Patients
Brief Title: Accessible Cancer Care to Enable Support for Survivors Programme
Acronym: ACCESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Singapore (Other)
Collaborators: National Cancer Centre, Singapore (Other)
Responsible Party: Principal Investigator, Alexandre Chan, Associate Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CIRB Ref. No: 2019/2090
Record Dates: First submitted 2019-07-04; First posted 2019-07-10 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Survivorship; Breast Cancer; Gynecologic Cancer
Keywords: distress screening; supportive care; survivorship; health service; triage; breast cancer; gynecologic Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: In this cluster randomized study, a cluster unit is defined as the clinic held by the individual oncologists who are treating eligible patients. The randomization schedule will allocate the cluster units (i.e. each oncologist and their clinic) in a 1:1 ratio to either the new supportive and survivorship care program or usual care arm. Therefore, all participants who received care from the same oncologist will have the same allocation.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supportive and survivorship care program (Experimental): Routine distress screening will be conducted using the Distress Thermometer (DT) and an accompanying problem list. Participants will complete the screening tool before their consults with oncologists and the results will be stored in their medical records. During the consult, oncologists will review the DT scores and problem list with each participant to provide the corresponding educational materials, advice or referrals. Highly distressed participants may be referred by oncologists to the supportive care nurses (SCN) for further triage and review.
  Interventions: Other: Supportive and survivorship care program
- Usual care (Placebo Comparator): No routine distress screening will be performed.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Supportive and survivorship care program — Provision of routine systematic screening using distress thermometer and problem list with accompanying supportive care nurse service.
  Arms: Supportive and survivorship care program
Other: Usual care — Usual care
  Arms: Usual care

SUMMARY:
In Singapore, cancer patients are not consistently assessed for unmet survivorship care needs and systematically identified for subsequent referral to useful care services. To address this gap, a preliminary multidisciplinary program is developed to (i) routinely screen and identify cancer patients with high distress levels, and (ii) provide appropriate care referrals after a systematic review by a supportive care nurse.

This study hypothesized that breast and gynecological cancer patients receiving timely screening for distress and appropriate supportive care services will report better improvement in quality of life as compared to non-recipients under usual care. This pilot study then aims to evaluate:

(i) The effectiveness of the program on a patient level in improving the quality of life and the symptom burden of patients requiring further supportive services.

(ii) The feasibility of the program's implementation on a health-system level among breast and gynaecological cancer patients in the outpatient oncology clinics at a specialty cancer centre.

DETAILED DESCRIPTION:
A cluster randomized controlled trial will be conducted at the National Cancer Centre Singapore (NCCS) over a period of 2 years. Eligible participants and their caregivers where applicable will be recruited and followed-up for a period of 12 months. Patients in the intervention arm will receive routine distress screening and referral to a supportive care nurse service where necessary; whereas patients in the control arm will receive usual care.

Patients' quality of life will be assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) and compared longitudinally between both study arms at a 3-months interval. Additionally, physical and psychological symptom distress levels will be compared using the Rotterdam Symptom Checklist (RSCL).

For patients who receive symptom-specific services, additional questionnaires will be completed before and after they have received the service. They include the following: Multi-dimensional Fatigue Symptom Inventory-Short Form (MFSI-SF) for fatigue, Patient Neurotoxicity Questionnaire (PNQ) for neuropathy, Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog v3.0) for cognitive function, and Patient-Reported Arthralgia Inventory (PRAI) for arthralgia.

An economic evaluation will be conducted using healthcare resource utilization and cost data gathered from health records and surveys including the Work Productivity and Activity Impairment (WPAI) questionnaire. Process outcomes of the program delivery will also be obtained to assess its feasibility by monitoring the referral patterns to supportive care nurse and adherence to screening or appointments. Lastly, patient satisfaction and clinicians acceptability of the program will be assessed via questionnaires.

Results from this study on the program's feasibility and effectiveness among breast and gynecological cancer patients are crucial to highlight potential implementation barriers and utility for patients before extending to other cancer types. Furthermore, results can shed a light on the program's scalability for future integration into routine care. This compelling initiative will contribute to the institution of integrated and coordinated rehabilitative and specialized clinics services to address supportive and survivorship needs of cancer patients across the continuum in the long run.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of breast or gynaecological cancer ascertained by clinical documentation
* Newly diagnosed patients receiving subsequent follow-up care in NCCS
* Able to read and understand English or Chinese
* Capable of providing informed consent

Exclusion Criteria:

* Physically or mentally incapable of providing verbal / written consent
* Patients under active care by the palliative care team

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life from baseline across all time points between the intervention and control study arm | Once at baseline and every 3 months for a period of 12 months
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ-C30) assesses cancer patients' health-related quality of life for the past week. The global quality of life status scale will be used and it is scored from 0 to 100 where a higher score is indicative of better functioning.

SECONDARY OUTCOMES:
Proportion of patients who achieve a clinically significant improvement or deterioration in quality of life between the intervention and control study arm | 12 months post recruitment
  Difference in quality of life scores assessed by EORTC QLQ-C30 will be tabulated for each patient. For each subscale, a medium improvement and deterioration in the longitudinal scores are defined and the proportion of patients who achieved the improvement or deterioration will be tabulated.
Physical and psychological symptom distress levels between the intervention and control study arm | Once at baseline and every 3 months for a period of 12 months
  The physical domain of the Rotterdam Symptom Checklist (RSCL) comprises of 23 items and the psychological distress domain comprises of 7 items. Patients will rate each item/ symptom on a 4-point Likert scale ("not at all", "a little", "quite a bit" and "very much"). A higher domain score indicates higher distress levels and symptom burden.
Quality of life of caregivers providing care to patients in the intervention study arm | 12 months post recruitment
  The Singapore Caregiver Quality of Life Scale (SCQOLS) is a validated, multi-domain quality of life measurement scale. The five domains consist of: physical well-being, mental well-being, experience and meaning, impact on daily living and financial well-being. A total QOL score will also be tabulated. A higher score in each domain and the total score will indicate better performance and quality of life respectively.
Fatigue levels | Baseline and 3 months after
  The Multi-dimensional Fatigue Symptom Inventory-Short Form (MSFI-SF) consists of 30 items to assess 5 dimensions of fatigue: physical, general, emotional, mental and vigour26. Respondent will rate each statement on a 5-point Likert scale from 0 ("not at all") to 4 ("extremely").
Severity of neuropathy | Baseline and 3 months after
  The Patient Neurotoxicity Questionnaire (PNQ) is a self-administered instrument designed for patient-based assessment of chemotherapy-induced peripheral neuropathy. It consists of two items that identify the incidence and severity of the sensory and motor disturbances. The severity will be rated from grade A to E with increasing severity. Also, patient will indicate the daily living activities that were interfered by chemotherapy treatment.
Cognitive function | Baseline and 3 months after
  The Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog v3.0) consists of 37 items to assess subjective cognitive function in the following 6 domains: memory, concentration, mental acuity, verbal fluency, functional interference and multitasking. Two other subscales included are "noticeability" of cognitive changes and "effect of perceived cognitive impairment on quality of life". Respondent will rate the frequency of occurrence of each item in the past week on a 5-point Likert scale from 0 ("never") to 4 ("several times a day"). A higher domain or subscale score indicating better perceived cognitive functioning.
Severity of arthralgia | Baseline and 3 months after
  The Patient-Reported Arthralgia Inventory (PRAI) consists of 16 items to measure arthralgia severity in 8 joint pair groups. Respondent will rate the pain severity at each joint for the past week using a 11-point Likert scale from 0 ("none") to 10 ("as bad as you can imagine"). The total score will be a sum of ratings for all items and range from 0 to 160 where a higher score indicates greater arthralgia severity.
Satisfaction levels of patients in the intervention study arm | 12 months post recruitment
  Patient acceptability questionnaire is adapted from the literature. Patients will rate the various processes in the program based on perceptions of the screening process, consult with supportive care nurse to discuss problems and the adequacy of information provision.
Work productivity | 9 months and 12 months post recruitment
  The Work Productivity and Activity Impairment (WPAI) questionnaire is a 6-item patient-reported quantitative assessment of the amount of absenteeism, presenteeism and daily activity impairment attributable to a specific health condition (cancer status) for the past week.
Extent of healthcare resource utilization | Throughout 12 months of follow-up period
  Information on outpatient visits, hospitalizations, and healthcare-related resources will be extracted from participants' medical and billing records.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Chan, PharmD, Principal Investigator — National University of Singapore, National Cancer Centre Singapore
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loh KW, Ng T, Choo SP, Saw HM, Mahendran R, Tan C, Chang GCY, Ong YJ, Yee ACP, Chan A, Soo KC. Cancer Supportive and Survivorship Care in Singapore: Current Challenges and Future Outlook. J Glob Oncol. 2018 Sep;4:1-8. doi: 10.1200/JGO.17.00117. PMID 30241247
- [Background] Tan ML, Idris DB, Teo LW, Loh SY, Seow GC, Chia YY, Tin AS. Validation of EORTC QLQ-C30 and QLQ-BR23 questionnaires in the measurement of quality of life of breast cancer patients in Singapore. Asia Pac J Oncol Nurs. 2014 Apr-Jun;1(1):22-32. doi: 10.4103/2347-5625.135817. PMID 27981079
- [Background] de Haes JC, van Knippenberg FC, Neijt JP. Measuring psychological and physical distress in cancer patients: structure and application of the Rotterdam Symptom Checklist. Br J Cancer. 1990 Dec;62(6):1034-8. doi: 10.1038/bjc.1990.434. PMID 2257209
- [Background] Lim HA, Mahendran R, Chua J, Peh CX, Lim SE, Kua EH. The Distress Thermometer as an ultra-short screening tool: a first validation study for mixed-cancer outpatients in Singapore. Compr Psychiatry. 2014 May;55(4):1055-62. doi: 10.1016/j.comppsych.2014.01.008. Epub 2014 Jan 18. PMID 24556515
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Cheung YB, Neo SHS, Teo I, Yang GM, Lee GL, Thumboo J, Chia JWK, Koh ARX, Qu DLM, Che WWL, Lau A, Wee HL. Development and evaluation of a quality of life measurement scale in English and Chinese for family caregivers of patients with advanced cancers. Health Qual Life Outcomes. 2019 Feb 14;17(1):35. doi: 10.1186/s12955-019-1108-y. PMID 30764839
- [Background] Reilly MC, Zbrozek AS, Dukes EM. The validity and reproducibility of a work productivity and activity impairment instrument. Pharmacoeconomics. 1993 Nov;4(5):353-65. doi: 10.2165/00019053-199304050-00006. PMID 10146874
- [Background] Chan A, Lew C, Wang XJ, Ng T, Chae JW, Yeo HL, Shwe M, Gan YX. Psychometric properties and measurement equivalence of the Multidimensional Fatigue Syndrome Inventory- Short Form (MFSI-SF) amongst breast cancer and lymphoma patients in Singapore. Health Qual Life Outcomes. 2018 Jan 19;16(1):20. doi: 10.1186/s12955-018-0846-6. PMID 29351803
- [Background] Kuroi K, Shimozuma K, Ohashi Y, Hisamatsu K, Masuda N, Takeuchi A, Aranishi T, Morita S, Ohsumi S, Hausheer FH. Prospective assessment of chemotherapy-induced peripheral neuropathy due to weekly paclitaxel in patients with advanced or metastatic breast cancer (CSP-HOR 02 study). Support Care Cancer. 2009 Aug;17(8):1071-80. doi: 10.1007/s00520-008-0550-x. Epub 2008 Dec 17. PMID 19089463
- [Background] Castel LD, Wallston KA, Saville BR, Alvarez JR, Shields BD, Feurer ID, Cella D. Validity and reliability of the Patient-Reported Arthralgia Inventory: validation of a newly-developed survey instrument to measure arthralgia. Patient Relat Outcome Meas. 2015 Jul 28;6:205-14. doi: 10.2147/PROM.S47997. eCollection 2015. PMID 26251635
- [Background] van Nuenen FM, Donofrio SM, Tuinman MA, van de Wiel HB, Hoekstra-Weebers JE. Feasibility of implementing the 'Screening for Distress and Referral Need' process in 23 Dutch hospitals. Support Care Cancer. 2017 Jan;25(1):103-110. doi: 10.1007/s00520-016-3387-8. Epub 2016 Aug 26. PMID 27565789
- [Background] Ristevski E, Regan M, Jones R, Breen S, Batson A, McGrail MR. Cancer patient and clinician acceptability and feasibility of a supportive care screening and referral process. Health Expect. 2015 Jun;18(3):406-18. doi: 10.1111/hex.12045. Epub 2013 Jan 31. PMID 23369083
- [Background] Cocks K, King MT, Velikova G, de Castro G Jr, Martyn St-James M, Fayers PM, Brown JM. Evidence-based guidelines for interpreting change scores for the European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30. Eur J Cancer. 2012 Jul;48(11):1713-21. doi: 10.1016/j.ejca.2012.02.059. Epub 2012 Mar 12. PMID 22418017